CLINICAL TRIAL: NCT05462158
Title: The Impact on Nudges of CKD Testing
Brief Title: Message Testing for CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 850936
Record Dates: First submitted 2022-04-24; First posted 2022-07-18 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Available for Members Text Message; Checked Health Text Message; No Text Message

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Available for Members-Text (Experimental): Participants will receive a text message that says, "Two common kidney tests have been made available for members. By taking them, you could stay ahead of any problems and keep enjoying life. Schedule a doctor visit today to ask about them.
  Interventions: Behavioral: Impact of Nudges on CKD Testing
- Checked Health-Text (Experimental): Participants will receive a text message that will say, "Have you checked your kidney health recently? By taking two common kidney tests, members can stay ahead of any problems and keep enjoying life. Schedule a doctor visit today to ask about them."
  Interventions: Behavioral: Impact of Nudges on CKD Testing
- No Text Message (Experimental): Participants in this group will not receive a text message at all
  Interventions: Behavioral: Impact of Nudges on CKD Testing

INTERVENTIONS:
Behavioral: Impact of Nudges on CKD Testing — The investigators will examine the impact of different messages on different dimensions of testing for CKD

SUMMARY:
Members of CVS/Aetna will receive one of two text messages or receive no text message at all. In the available for members condition, participants will receive a text message that says, "Two common kidney tests have been made available for members. By taking them, you could stay ahead of any problems and keep enjoying life. Schedule a doctor visit today to ask about them." In the Checked Health condition, the message will say, "Have you checked your kidney health recently? By taking two common kidney tests, members can stay ahead of any problems and keep enjoying life. Schedule a doctor visit today to ask about them." There will also be a group of members that do not receive a text message at all.

DETAILED DESCRIPTION:
The investigators will examine the proportion of participants that book an appointment, proportion of new diagnoses for CKD, creatinine tests and/or albuminuria tests, proportion of participants that looked for more information after receiving the text message. The investigators will examine these metrics 6 months after all of the text messages have gone out ~8,637. The investigators will examine difference in conditions between the metrics listed above in the DV section. The investigators will compare the two conditions to each other, as well as to the group who does not receive a text message. The investigators will conduct a series of chi square tests/logistic regressions to examine the differences.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a health insurance customer with the company we are working with.
* All other eligibility criteria are determined by the company and not disclosed to us. They will pick a sample of customers for the study, with participants then being randomly assigned to treatments they qualify for.

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8637 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Proportion of appointments | The investigators will examine this 6 months after all of the text messages are sent out~8637 of them
  The investigators will examine the proportion of appointments participants make between conditions
Proportion of new diagnoses for CKD, creatinine tests and/or albuminuria tests | The investigators will examine this 6 months after all of the text messages are sent out~8637 of them
Proportion of participants that looked for more information | The investigators will examine this 6 months after all of the text messages are sent out~8637 of them
  Participants can request for more information upon receiving the text message

CONTACTS AND LOCATIONS:
Overall Officials: Marissa Sharif, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Health Incentives and Behavioral Economics (CHIBE), Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
The company we are working with will be analyzing the data and informing us of the results. We will not have data to share.